CLINICAL TRIAL: NCT02782832
Title: No Need for Neuromuscular Blockade in Day Case Standardised Laparoscopic Surgery. A Consecutive Retrospective Study
Brief Title: No Need for Neuromuscular Blockade in Daycase Laparoscopic Surgery
Status: Completed | Type: Observational
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Billy B Kristensen, Chief Physician, Hvidovre University Hospital
Other Study IDs: DagKir-neuromus block
Record Dates: First submitted 2016-02-15; First posted 2016-05-25 (Estimated); Last update posted 2018-05-29 (Actual); Status verified 2018-05

CONDITIONS: Cholecystitis; Inguinal Hernia, Direct; Umbilical Hernia
Keywords: Neuromuscular; Blockade; Surgery
MeSH Terms: conditions — Cholecystitis; Hernia, Inguinal; Hernia, Umbilical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study analyse the need for neuromuscular blockade in consecutive routine laparoscopic procedures without standard use of neuromuscular blockade in an ambulatory laparoscopic surgery setting and analyse specific reasons for using neuromuscular blockade in individual patients. Furthermore, the study report the analgesic use in postoperative care unit and the discharge rate.

DETAILED DESCRIPTION:
The study is retrospective, including consecutive patients in an unrestricted referral of patients undergoing laparoscopic cholecystectomy, umbilical and inguinal hernia repair. Inclusion period was from 01.04.2013 to 31.03.2015. All patients received general anesthesia using propofol (2 mg/kg) and remifentanil (1 μg/kg/min) for induction. In patients where tracheal intubation was required, this was done without use of neuromuscular blocking drug; otherwise a proseal laryngeal mask was used. For the maintenance of anesthesia, additional continuous infusion of propofol (3-5 mg/kg/h) and remifentanil (0.3-0.5 μg/kg/min) was used. Data were derived from a prospective local database on demographics, anesthetic methods and supplements (i.e. need for neuromuscular blockade) and postoperative needs for supplementary analgesics besides the postoperative standard analgesic regimen, number of hours stayed in the ambulatory surgery department, and discharge rate (including reasons for hospital admittance).

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing laparoscopic cholecystectomy, umbilical and inguinal hernia repair

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Retrospective study, including consecutive patients in an unrestricted referral of patients undergoing laparoscopic cholecystectomy, umbilical and inguinal hernia repair
Sampling Method: Probability Sample
Enrollment: 1245 (Actual)
Dates: Start 2016-05; Primary Completion 2016-06 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Number of patients requiring neuromuscular blockade | At time of surgery
  Data derived from a prospective local database on need for neuromuscular blockade in patients undergoing laparoscopic cholecystectomy, umbilical and inguinal hernia repair.

SECONDARY OUTCOMES:
Analgesic use in postoperative care unit | Within 6 hours after surgery
  Amount of opioids administered to the patients in the postoperative care unit
Hours stayed in the postoperative care unit | 1 to 6 hours after surgery
Maximum Visual analog score (VAS) for pain in the postoperative Care unit | 1 to 6 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Billy B Kristensen, MD, Principal Investigator — Hvidovre University Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Staehr-Rye AK, Rasmussen LS, Rosenberg J, Juul P, Lindekaer AL, Riber C, Gatke MR. Surgical space conditions during low-pressure laparoscopic cholecystectomy with deep versus moderate neuromuscular blockade: a randomized clinical study. Anesth Analg. 2014 Nov;119(5):1084-92. doi: 10.1213/ANE.0000000000000316. PMID 24977638
- [Background] Staehr-Rye AK, Rasmussen LS, Rosenberg J, Juul P, Gatke MR. Optimized surgical space during low-pressure laparoscopy with deep neuromuscular blockade. Dan Med J. 2013 Feb;60(2):A4579. PMID 23461992
- [Background] Martini CH, Boon M, Bevers RF, Aarts LP, Dahan A. Evaluation of surgical conditions during laparoscopic surgery in patients with moderate vs deep neuromuscular block. Br J Anaesth. 2014 Mar;112(3):498-505. doi: 10.1093/bja/aet377. Epub 2013 Nov 15. PMID 24240315
- [Background] Kopman AF, Naguib M. Laparoscopic surgery and muscle relaxants: is deep block helpful? Anesth Analg. 2015 Jan;120(1):51-58. doi: 10.1213/ANE.0000000000000471. PMID 25625254
- [Background] Abrishami A, Ho J, Wong J, Yin L, Chung F. Sugammadex, a selective reversal medication for preventing postoperative residual neuromuscular blockade. Cochrane Database Syst Rev. 2009 Oct 7;(4):CD007362. doi: 10.1002/14651858.CD007362.pub2. PMID 19821409
- [Background] Barczynski M, Herman RM. A prospective randomized trial on comparison of low-pressure (LP) and standard-pressure (SP) pneumoperitoneum for laparoscopic cholecystectomy. Surg Endosc. 2003 Apr;17(4):533-8. doi: 10.1007/s00464-002-9121-2. Epub 2003 Feb 17. PMID 12582754
- [Background] Wallace DH, Serpell MG, Baxter JN, O'Dwyer PJ. Randomized trial of different insufflation pressures for laparoscopic cholecystectomy. Br J Surg. 1997 Apr;84(4):455-8. PMID 9112891
- [Background] Perrakis E, Vezakis A, Velimezis G, Savanis G, Deverakis S, Antoniades J, Sagkana E. Randomized comparison between different insufflation pressures for laparoscopic cholecystectomy. Surg Laparosc Endosc Percutan Tech. 2003 Aug;13(4):245-9. doi: 10.1097/00129689-200308000-00004. PMID 12960786
- [Background] Larsen JF, Ejstrud P, Kristensen JU, Svendsen F, Redke F, Pedersen V. Randomized comparison of conventional and gasless laparoscopic cholecystectomy: operative technique, postoperative course, and recovery. J Gastrointest Surg. 2001 May-Jun;5(3):330-5. doi: 10.1016/s1091-255x(01)80056-1. PMID 11360058
- [Derived] Loven H, Kristensen BB, Bisgaard T. Low admittance rate after ambulatory laparoscopic surgery. Dan Med J. 2019 Jun;66(6):A5547. PMID 31256774